CLINICAL TRIAL: NCT07145086
Title: Translaryngeal Vibration for Hyperfunctional Voice Disorders
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Christian University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R15DC021255-01A1 (NIH); 1R15DC021255-01A1 (NIH)
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Dysphonia; Muscle Tension Dysphonia
Keywords: Dysphonia; Muscle Tension Dysphonia; Voice Therapy; Vibration
MeSH Terms: conditions — Dysphonia | interventions — Vibration

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Five Week Therapy (Experimental): Participants receive five weeks of voice therapy with vibration
  Interventions: Behavioral: Voice therapy with vibration
- Eight Week Therapy (Active Comparator): Participants receive eight weeks of voice therapy with vibration
  Interventions: Behavioral: Voice therapy with vibration
- Voice Therapy with Placebo (Placebo Comparator): Participants receive eight weeks of voice therapy with vibration placebo
  Interventions: Behavioral: Voice therapy with vibration

INTERVENTIONS:
Behavioral: Voice therapy with vibration — Voice therapy with a novel vibration device will be delivered for five or eight weeks depending on group allocation. All participants will receive flow phonation voice therapy.

SUMMARY:
Contemporary treatments for hyperfunctional voice disorders such as muscle tension dysphonia (MTD) are effective but typically do not restore voice handicap or voice function to normal thresholds. Recent reports of vibration as a voice therapy modality have been published, but many questions remain about the efficacy of this tool. The current project addresses these problems through a blinded and randomized controlled trial to investigate the efficacy of local translaryngeal vibration for MTD and the dose-response relationship of this modality when compared to treatment without vibration.

DETAILED DESCRIPTION:
High-quality research designs have demonstrated that voice therapy has a positive impact on hyperfunctional voice disorders associated with muscle tension dysphonia (MTD). Among the options of behavioral voice therapy for MTD, one of the most effective evidence-based approaches is flow phonation (a.k.a., stretch-and-flow voice therapy). However, the phenomenon of post-treatment outcome measures remaining substantially outside the range of normal is a ubiquitous finding in studies investigating this and other voice therapy approaches. From both a cost burden and quality of life perspective, this phenomenon supports a need to develop and refine voice therapy treatment approaches to promote better outcomes. Vibration is a physical modality that has a historical use in the rehabilitation professions, but only recently has it been scientifically studied as a modality for voice therapy when used by speech-language pathologists. When applied locally on the perilaryngeal surface as a local translaryngeal vibration therapy (LTLV), early research has demonstrated beneficial effects on voice physiology and clinical outcomes. Further high-quality clinical research studies are needed to evaluate the efficacy of LTLV as a modality for voice disorders and to better understand the effects of vibration and effective vibration dose on voice rehabilitation outcomes. The research proposed in this R15 has the potential to transform clinical practice of treatment for MTD, the most common voice disorder among treatment-seeking populations. That potential is vested in the pursuit of three specific aims: (1) determine the clinical efficacy of LTLV as a concurrent treatment using flow phonation voice therapy in patients with MTD, and (2) determine the effect of treatment dose on clinical response associated with treatment outcomes. In addition to the potential impact of this R15, the innovative of approach of using LTLV as a concurrent modality with flow phonation combined with investigation of the most effective frequency parameter for clinical application represents a pioneering approach to advance the field of clinical voice practice in speech-language pathology.

ELIGIBILITY:
Inclusion Criteria:

* a) diagnosis by an otolaryngologist of hyperfunctional dysphonia (MTD) without benign mid-membranous lesion (i.e., primary MTD or non-phonotraumatic hyperfunction) with and a recommendation for voice therapy, ((b) confirmation of dysphonia by a comprehensive voice evaluation conducted by a speech-language pathologist with experience in the evaluation and treatment of voice disordered populations, (c) to prevent floor effects of our primary outcome variable, participants will be required to exhibit a pre-treatment VHI score of >20, as this is the upper range for normal cutoff values in studies which have demonstrated high sensitivity and specificity for this tool (Behlau et al., 2016), (d) 18 years of age or older, (e) no history of local vibration therapy as part of a rehabilitation treatment program.

Exclusion Criteria:

* Unable to receive vibration to neck area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Voice Handicap Index | From enrollment to the end of treatment at 5 or 8 weeks"
  The Voice Handicap Index (VHI) is a self-assessment tool used to evaluate how a voice disorder impacts a person's daily life, encompassing functional, physical, and emotional aspects. It helps quantify the perceived handicap caused by a voice problem, aiding in diagnosis, treatment planning, and assessing treatment effectiveness. The VHI consists of 30 questions, divided into three subscales, with scores ranging from 0 to 120, where higher scores indicate a greater perceived handicap

SECONDARY OUTCOMES:
Consensus Auditory-Perceptual Evaluation of Voice | From enrollment to the end of treatment at 5 or 8 weeks"
  Perceptual Voice Quality measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No